CLINICAL TRIAL: NCT05459246
Title: The Effect of Virtual Reality Application on Pain Severity, Anxiety Level and Patient Satisfaction in Patients Who Will Be Applied Coronary Angiography
Brief Title: The Effect of Virtual Reality Application on Pain Severity, Anxiety Level and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Principal Investigator, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6811
Record Dates: First submitted 2022-07-06; First posted 2022-07-14 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Anxiety; Pain
Keywords: virtual reality glasses; Pain; Anxiety; Angiography.
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Virtual reality glasses and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality glasses (Experimental): Beginning 1 minute before the start of the procedure, the patients will be watched (30-45 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product "Secret Garden", during the procedure (30-45 minutes).
  Interventions: Other: Virtual reality glasses
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Virtual reality glasses — Beginning 1 minute before the start of the procedure, the patients will be watched (30-45 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product "Secret Garden", during the procedure (30-45 minutes).
  Arms: Virtual reality glasses

SUMMARY:
In this study; It is aimed to examine the Effect of Virtual Reality Based Relaxation Program on Pain Severity, Anxiety Level and Patient Satisfaction in Patients Who Will Be Applied Angiography.

DETAILED DESCRIPTION:
Beginning 1 minute before the start of the procedure, the patients will be watched (30-45 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product "Secret Garden", during the procedure (30-45 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Ability to communicate adequately
* Absence of psychiatric problems
* Volunteering to participate in the research
* Experiencing coronary angiography for the first time

Exclusion Criteria:

* Those who have communication problems
* Those with psychiatric problems
* Emergency coronary angiography
* Having symptoms of myocardial infarction,
* Being unconscious,
* Having surgery in the last 6 weeks,

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Before angiography (mean 6 months after study completion)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Visual Analog Scale | After angiography (through study completion, an average of 6 month)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Anxiety Assessment Scale | Before angiography (mean 6 months after study completion)
  Patients will be asked to show their anxiety levels before and after the procedure on a 10 cm long horizontal line. Line has 0 at the beginning and 10 at the end. 10 means very extreme anxiety and 0 means no anxiety.
Anxiety Assessment Scale | After angiography (through study completion, an average of 6 month)
  Patients will be asked to show their anxiety levels before and after the procedure on a 10 cm long horizontal line. Line has 0 at the beginning and 10 at the end. 10 means very extreme anxiety and 0 means no anxiety.
Physiological Symptoms of Anxiety Follow-up Form | Before angiography (mean 6 months after study completion)
  This form was created by the researcher to record blood pressure, heart rate, respiratory rate and peripheral oxygen saturation (SpO2) value.
Physiological Symptoms of Anxiety Follow-up Form | After angiography (through study completion, an average of 6 month)
  This form was created by the researcher to record blood pressure, heart rate, respiratory rate and peripheral oxygen saturation (SpO2) value.
Virtual Reality Glasses Application Satisfaction Form | Before angiography (mean 6 months after study completion)
  In this form, there are questions prepared in line with the relevant literature in order to determine the satisfaction with the video watched with virtual reality glasses.
Virtual Reality Glasses Application Satisfaction Form | After angiography (through study completion, an average of 6 month)
  In this form, there are questions prepared in line with the relevant literature in order to determine the satisfaction with the video watched with virtual reality glasses.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, PhD, Study Chair — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Güneydoğu Anadolu Bölgesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973